CLINICAL TRIAL: NCT05163535
Title: Open Labelled, Randomized Study to Evaluate the Efficacy, Safety and Dose Selection of VM-1500A-LAI Drug in HIV-infected Patients Transferred From Previous Stable Therapy (NNRTI + 2NRTI), Including ELPIDA®
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Viriom (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIV-VM1500ALAI-02
Record Dates: First submitted 2021-12-06; First posted 2021-12-20 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: HIV-1-infection
Keywords: HIV-1; LAI
MeSH Terms: interventions — elsulfavirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- VM-1500A-LAI (1200 mg, 1200 mg, 1200 mg) (Experimental): VM-1500A-LAI 3 i / m injections with an interval of 4 weeks (1200 mg, 1200 mg, 1200 mg) during daily therapy with 2NRTIs for 12 weeks
  Interventions: Drug: VM-1500A-LAI
- VM-1500A-LAI (1200 mg, 900 mg, 900 mg) (Experimental): VM-1500A-LAI 3 i / m injections with an interval of 4 weeks (1200 mg, 900 mg, 900 mg) during daily therapy with 2NRTIs for 12 weeks
  Interventions: Drug: VM-1500A-LAI
- VM-1500A-LAI (1200 mg, 600 mg, 600 mg) (Experimental): VM-1500A-LAI 3 i / m injections with an interval of 4 weeks (1200 mg, 600 mg, 600 mg) during daily therapy with 2NRTIs for 12 weeks
  Interventions: Drug: VM-1500A-LAI
- ELPIDA® (Other): ELPIDA®, 20 mg capsules and 2NRTIs, daily therapy for 12 weeks
  Interventions: Other: ELPIDA®

INTERVENTIONS:
Drug: VM-1500A-LAI — VM-1500A (parent drug of elsulfavirine) IM injection dosage form
  Other Names: VM-1500A; VM-1500; ELPIDA®
  Arms: VM-1500A-LAI (1200 mg, 1200 mg, 1200 mg); VM-1500A-LAI (1200 mg, 600 mg, 600 mg); VM-1500A-LAI (1200 mg, 900 mg, 900 mg)
Other: ELPIDA® — Elsulfavirine capsules
  Other Names: VM-1500
  Arms: ELPIDA®

SUMMARY:
Open labelled, randomized study to evaluate the efficacy, safety and dose selection of VM-1500A-LAI drug in HIV-infected patients transferred from previous stable therapy (NNRTI + 2NRTI), including ELPIDA®.

DETAILED DESCRIPTION:
The clinical study will consist of the following stages:

1. Screening:

   On Week 2, after signing the Patient Information Sheet and the Informed Consent form, subjects will undergo screening procedures to assess the inclusion/exclusion criteria. Patients meeting all inclusion / exclusion criteria will be invited to the center for randomization and initiation of study drug therapy.
2. Study treatment period:

   Once the inclusion / exclusion criteria have been confirmed, patients will be randomized to one of four treatment groups. For patients assigned to Groups 1, 2 and 3, all i/m injections of VM-1500A-LAI will be administered at Week 0, Week 4 and Week 8 by the study physician at the center, where they will remain monitored for up to 2 hours. Patients will also receive 2NRTI according to the standard regimen. Blood samples for PK study will be taken immediately before and 2 hours after each i/m injection of VM-1500A-LAI. Patients assigned to Group 4 will receive daily ELPIDA® 20 mg in the morning and 2NRTIs according to the standard regimen.
3. End of Therapy:

   At the end of the study therapy course, patients will be invited to the study center for a Week 12 visit for the end of therapy visit procedures.
4. Follow-up Observation period:

After the end of the course of study therapy, patients will be monitored for another 4 weeks. Patients will be invited to the center for a Follow-up Visit at Week 16. Follow-Up to obtain the data on adverse events will be continued for up to 30 days after the last visit or the last study procedure planned in the Study Protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Patient Information Sheet and Informed Consent Form
2. Men and women aged 18 and over;
3. HIV-1 infection confirmed serologically by ELISA or immunoblot analysis (or documented HIV-1 infection);
4. Clinically stable HIV infection (clinical stages 1 or 2 according to the WHO classification, Appendix 1)
5. Stable doses of NNRTIs (ELPIDA®, 20 mg capsules) + 2NRTIs for 6 months before screening;
6. HIV-1 RNA plasma level ≤ 50 copies/ml at screening;
7. СD4+ Т-cells count ≥ 200 cells/mm3 at screening;
8. Laboratory parameters;
9. The patients' consent to use adequate contraception methods during the study (condom with spermicide).

Exclusion Criteria:

1. Presence of known primary HIV-1 resistance to ART. Viral resistance mutations are defined as any basic mutations of resistance to NNRTI pursuant to the renewed list of the International Community of HIV-1 Resistant AIDS Mutations (2013) associated with drug resistance for any genotype.
2. Acute hepatitis or cirrhosis of the liver of any etiology; HBsAg or antibodies to hepatitis C (in the case of Anti-HCV +, the exclusion criterion must be confirmed by determining a positive HCV RNA test) at screening;
3. Signs of acute infection or presence of syphilis, hepatitis A, Toxoplasma gondii, cytomegalovirus, gonorrhea and Chlamydia trachomatis tests results within 30 days prior to screening
4. Opportunistic infections referred to Category C of the classification of the Center for disease control (CDC), dated 2008, except for Kaposi's sarcoma not requiring system therapy;
5. History of tuberculosis of any localization or on screening according to chest x-ray (in frontal and lateral projections);
6. History of malignant neoplasms (except for basal cell epithelioma or squamous cell carcinoma of skin and in situ cervical carcinoma, which were resected and healed more than 5 years ago);
7. Participation in other clinical studies or therapy with other study drugs within 3 months before Screening. Patients who participated in study HIV-VM1500-06 may be included in this study;
8. Course intake of immunomodulators (interferons, interleukins), immune-suppresive therapy (cyclosporins), glucocorticoids 1 month before screening
9. Current alcoholic or drug addiction, which the researcher may think to hinder the patient to take part in the study and adhere to all requirements per protocol
10. Hypersensitivity to any component of the study drug; hypersensitivity to any of the components, including lactose intolerance, or the presence of contraindications to the appointment of ELPIDA® or ART drugs;
11. Taking excluded drugs from the list of "excluded drugs";
12. Taking other study drugs for 12 weeks or 5 drug half-lives (whichever is longer) prior to screening;
13. Signs of expressed uncontrolled associated disease, e.g., disorders of nervous, respiratory, cardiac-vessel (including unstable angina, myocardial infarction, transient ischemic attack or stroke 12 months before screening) systems, kidneys, liver, endocrinic system and gastrointestinal tract, which as the Investigator may think could prevent the patient from participation in the study;
14. Systemic autoimmune disorders and connective tissue diseases, which require prior or current treatment with systemic glucocorticoid drugs, cytostatics or penicillamine;
15. Pregnant or lactating women or women planning to get pregnant during the clinical study; women at the child-birthing age (including non-sterilized by surgical means during post-menopause period less than 2 years), who do not use adequate contraception methods;
16. Inability to read or write; unwillingness to understand and adhere to the study protocol procedures; non-compliance with the drugs intake regimen or execution of procedures, which as the Investigator believes may affect the study results or subject's safety and prevent the subject from further participation in the study; any other concomitant medical or serious psychological conditions making the subject not eligible to participate in the clinical study restrict the legality of obtaining the Informed Consent or may affect the patient's ability to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2021-08-03 (Actual); Study Completion 2021-08-03 (Actual)

PRIMARY OUTCOMES:
Concentration of VM1500A in plasma and RBCs | 16 weeks
  Assess the clinical and virological efficacy of three dosage regimens of VM-1500A-LAI in HIV-infected patients transferred to VM-1500A-LAI from previous stable therapy (NNRTI + 2NRTI), including ELPIDA®, 20 mg capsules, lasting at least 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Anastasia Pokrovskaya, PhD, Principal Investigator — Central Research Institute of Epidemiology of Rospotrebnadzor
Locations (2):
- Russia (2):
  - Federal State Budgetary Institution of the Central Research Institute of Epidemiology of Rospotrebnadzor, Moscow
  - St. Petersburg State Medical Institution " Center for AIDS and Infectious Diseases", Saint Petersburg

IPD SHARING:
Plan to Share IPD: No